CLINICAL TRIAL: NCT04761718
Title: Covid-19 Epidemic Lockdown Impact on Psychomotor Performance in Egyptian Children
Brief Title: Covid-19 Epidemic Lockdown Impact on Psychomotor Performance
Status: Completed | Type: Observational
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Amira Hussin Hussin Mohammed, Assistant. Professor of physical therapy, Department of Physical Therapy for Pediatrics, Delta University for Science and Technology
Other Study IDs: Covid-19 Epidemic impact
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Covid19 Epidemic Lockdown Impact

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
PURPOSE:

To detect the Covid-19 Epidemic Lockdown impact on Psychomotor performance in Egyptian Children.

BACKGROUND:

The corona virus disease (COVID-19) affected virtually all countries including Egypt as records showed 156,397 subjects including all age groups, Adolescents and children represent sector in the records, lockdown can contribute to widespread psychological distress and an increased risk of physical inactivity consequences shortly. Psychomotor disorders are expected during and aftermath of the pandemic. Validated Questionnaires are tools to assess the psychomotor condition during and after pandemic lockdown as safe and valid assessment tool.

HYPOTHESES:

Covid-19 Epidemic Lockdown has an impact on Psychomotor performance in Egyptian Children.

RESEARCH QUESTION:

Does Covid-19 Epidemic Lockdown impact on Psychomotor performance in Egyptian Children?

ELIGIBILITY:
Inclusion Criteria:

100 participants will be chosen according to the following criteria : subject in both sexes and their age will ranged between

1. 6-9 years.
2. 10-13 years.
3. 14-18 years All subjects should be clinically and medically stable

Exclusion Criteria:

Subjects with psychological or Motor impairment will be excluded from the study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants will be randomly selected from all provinces in Egypt.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2022-06-25 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
pre lockdown assessment for physical activity | up to 24 weeks
  Google form questionnaires include the physical activity questionnaire.
post lockdown assessment for physical activity | up to 24 weeks
  Google form questionnaires include the physical activity questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- AAA, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 12 months after publishing